CLINICAL TRIAL: NCT05619939
Title: Determining the Effect of Dietary Protein Source on Intestinal Health
Brief Title: Impact of Protein Source on Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Montrose, Principal Investigator, Stony Brook University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2022-00427
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Intervention Model Description: This study is designed as a single-blinded randomized crossover trial in which individuals will be assigned to 2 groups. One group will receive 10 days of pea protein isolate followed by 10 days of consuming egg white protein isolate, with the two treatment periods separated by a 14-day washout period. The second group will receive the isolates in the opposite order.
Who Masked: Participant
Masking Description: Subjects will be blinded as to which protein type they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pea protein to egg white protein (Experimental): This arm will receive 10 days of pea protein isolate followed by 10 days of consuming egg white protein isolate, with the two treatment periods separated by a 14-day washout period.
  Interventions: Dietary Supplement: Protein isolate
- Egg white protein to pea protein (Experimental): This arm will receive 10 days of egg white protein isolate followed by 10 days of consuming pea protein isolate, with the two treatment periods separated by a 14-day washout period.
  Interventions: Dietary Supplement: Protein isolate

INTERVENTIONS:
Dietary Supplement: Protein isolate — The indicated protein isolates will be given to subjects as their major protein source

SUMMARY:
The gastrointestinal (GI) tract is a central hub for human health given its essential role in nutrient absorption, waste production and immunity. Diet is a major contributor to gut health including affecting the incidence and severity of GI disease. This is mediated, at least in part, by the presence of microbiota, a highly diet-dependent biome. In fact, dietary changes are capable of altering bacterial populations and/or microbial metabolism, which in turn, controls the type and abundance of small molecules being produced in the gut, many of which can exert biological effects. Several lines of evidence suggest that dietary protein in particular, can impact gut health. Therefore, this trial will test whether dietary protein type differentially impacts gut function in humans by carrying out a single-blinded randomized cross-over controlled feeding study in healthy individuals. Subjects will be provided with an individualized very low protein diet augmented with pea- or egg white-derived protein supplements, as their major protein source. The impact of consuming pea vs. egg white protein on 1) the fecal metabolome, 2) gut barrier function and 3) gastrointestinal symptoms will be determined.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18-29.9

Exclusion Criteria:

* Those with a history of significant illness including diabetes, renal, liver or cardiovascular disease, malnutrition, GI disease (including IBS, IBD, chronic constipation or diarrhea), mental illness (i.e. depression, bipolar disorder)
* Those adhering to a vegan diet or vegetarian diet exclusive of eggs
* Those having taken probiotics or antibiotics within 1 month of starting the study
* Those who are pregnant or plan to become pregnant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Fecal metabolome | This analysis will be carried out at baseline and the end of each treatment period, entailing 4 measurements over an approximately 36 day period
  Mass-spectrometry based analysis of the relative abundance of metabolites will be carried out on feces.
Intestinal permeability | This analysis will be carried out at baseline and the end of each treatment period, entailing 4 measurements over an approximately 36 day period
  Subjects will undergo lactulose-mannitol test to inform on gut permeability

SECONDARY OUTCOMES:
Adherence to study diets | Daily over two, 10-day periods
  consumption of study diets will be recorded through subject-reported surveys before and after eating.
Amount of study diets consumed | Daily over two, 10-day periods
  Subjects will take pictures of food items before and after eating to assess the amount of each study diet item consumed.

CONTACTS AND LOCATIONS:
Overall Officials: David C Montrose, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States